CLINICAL TRIAL: NCT06317753
Title: Can Exercise Rewire the Brain Addiction Circuitry? A Randomized Trial of Exercise and Binge Drinking
Brief Title: Can Exercise Rewire the Brain Addiction Circuitry?
Acronym: REWIRED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Sonia Sousa, Principal Investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMinho1
Record Dates: First submitted 2024-03-02; First posted 2024-03-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Physical Exercise
Keywords: Addiction circuitry; Binge drinking; Neuroimaging
MeSH Terms: conditions — Motor Activity; Binge Drinking | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The protocol includes a randomized controlled trial with a follow-up at three months involving three groups of adolescents (18-24 Y) -experimental group 1, will be enrolled in the Aerobic program, experimental group 2 will be involved in the agility program, and an active control group that will be participating in a stretching program. Participants will be randomly assigned to each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental condition 1 (Experimental): Participants allocated to the Experimental condition 1 will be following a aerobic exercise training program.
  Interventions: Behavioral: Aerobic Exercise
- Experimental condition 2 (Experimental): Participants allocated to the Experimental condition 2 will be following an agility-cognitive exercise training program.
  Interventions: Behavioral: Agility-Cognitive Exercise
- Control condition (Active Comparator): Participants allocated to the Control condition will be following a stretching/relaxation training program.
  Interventions: Behavioral: Stretching/relaxation

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants allocated to the Aerobic condition will be following a 4 month-intervention aerobic exercise protocol of 3 weekly interleaved sessions with a 50 minutes duration
  Arms: Experimental condition 1
Behavioral: Agility-Cognitive Exercise — Participants allocated to the Agility-Cognitive condition will be following a 4 month-intervention agility-cognitive exercise protocol of 3 weekly interleaved sessions with a 50 minutes duration
  Arms: Experimental condition 2
Behavioral: Stretching/relaxation — Participants allocated to the stretching control condition will be following a 4 month-intervention protocol of 1 weekly session with a 50 minutes duration
  Arms: Control condition

SUMMARY:
The aim of the present study is to apply neuroimaging techniques to investigate how physical exercise may influence the addiction circuitry, ultimately reducing alcohol consumption and craving in youth binge drinkers. This proposal will advance knowledge on how exercise may modulate the neurocircuitry of addiction. Uncovering the neurobiological mechanisms underlying the interactive neural effects of exercise and alcohol intake may provide additional scientific insights for the development of preventive and intervention programs for youth BD and AUD.

DETAILED DESCRIPTION:
The proposed research plan focuses on the identification of changes in the structural and functional brain parameters (e.g. volume, brain activity), in response to a physical exercise (PE) protocol, on the neurocircuitry of addiction, after a 4 month-intervention program in college binge drinkers (BDs). The main objectives of this proposal are: O1) to evaluate the potential benefits of PE on the brain structure and function, particularly in the neurocircuitry of addiction, in a sample of Portuguese college students with a binge drinking pattern of alcohol use; and O2) to determine whether the PE intervention reduces craving and alcohol consumption levels in BDs. The present project will involve: i) a pre-intervention comprehensive evaluation of behavioral (alcohol consumption), psychological (craving levels), physiological (VO2, HRV), and neurological (neuroimaging) variables; ii) a training phase consisting of 48 sessions (3 weekly sessions*16 weeks) of aerobic (exp group 1), agility-cognitive (exp group 2) exercise and stretching (control group; iii) a post-intervention evaluation of behavioral, physiological, and neurological (neuroimaging) variables; iv) and a 6 months' follow- up evaluation of behavioral, physiologicaln and cognitive variables. A randomized controlled trial will be implemented at the University of Minho. It will include a total of 60 college students with a binge drinking pattern of alcohol intake, 20 participants per condition.

ELIGIBILITY:
Inclusion Criteria:

* binge drinking > or = 5 ; > or =4 for women alcoholic drinks
* in the same time window (±2h)
* at least once per month
* <150 minutes of physical activity per week

Exclusion Criteria:

* Major and/or unstable medical conditions
* Physical limitations that may constraint the practice of exercise
* Cardiovascular and respiratory insufficiency
* History of traumatic brain injury or neurological disorder
* Non-corrected sensory deficits
* Personal history of psychopathological disorders
* Family history of alcoholism or substance abuse in first degree relatives
* Consumption of medical drugs with psychoactive effects (e.g., sedatives or anxiolytics) during the month previous to the assessment
* Use of illegal drugs and AUDIT scores >20
* MRI contraindications
* Current or previous (past year) participation in a physical exercise program

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 50% male, 50% female
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Behavioral: alcohol consumption | Through study completion, an average of 1 year
  Number of drinks per binge drinking episode
Behavioral: binge episodes | Through study completion, an average of 1 year
  Number of binge drinking episodes
Behavioral : drunkenness | Through study completion, an average of 1 year
  Percentage of drunkenness
Psychological (craving levels) | Through study completion, an average of 1 year
  Scores in the Alcohol Craving Questionnaire (The cutoff points for total scale points are: 12-17 = minimal desire, 18-25 = mild, 26-42 = moderate and 43 or more = severe)
Brain structure | Through study completion, an average of 1 year
  Structure-volume in liters
Brain structural connectivity- FA | Through study completion, an average of 1 year
  Structural connectivity-fractional anisotropy-scalar value between zero and one within a voxel that describes the degree of anisotropy of a diffusion process
Brain structural connectivity - MD | Through study completion, an average of 1 year
  Structural connectivity-mean diffusivity-a scalar measure between zero and one that describes the total diffusion within a voxel
Brain structural connectivity - AD | Through study completion, an average of 1 year
  Structural connectivity-axial diffusivity-a scalar measure between zero and one within a voxel that describes the magnitude of diffusion parallel to fiber tracts.
Brain structural connectivity - RD | Through study completion, an average of 1 year
  Structural connectivity-radial diffusivity-a scalar measure between zero and one within a voxel that describes the magnitude of diffusion parallel to fiber tracts.
Brain function | Through study completion, an average of 1 year
  Bold signal for Task-related fMRI
Brain function-resting state | Through study completion, an average of 1 year
  Functional connectivity for resting-state fMRI

SECONDARY OUTCOMES:
Monetary Incentive Delay Task (included in the fMRI paradigm) - hits | Through study completion, an average of 1 year
  Accuracy, measured through the number of hits to assess the hypothetical differences in participant's level of achievement between the pretest, posttest and follow-up assessments.
Monetary Incentive Delay Task (included in the fMRI paradigm) - reaction time | Through study completion, an average of 1 year
  Reaction times, measured as seconds needed to give a response to assess the hypothetical differences in participant's level of achievement between the pretest, posttest and follow-up assessments.
Maximal oxygen consumption (VO2max) | Through study completion, an average of 1 year
  VO2max (ml/kg/min) will be measured in the pretest and posttest evaluations to assess the effects of the physical exercise protocol on cardiovascular fitness.
Brain-derived neurotrophic factor (BDNF) | Through study completion, an average of 1 year
  BDNF (pg/ml) concentrations measured in saliva will be measured in pre-intervention, post-intervention, at the midpoint of the intervention (2 months), and at the follow-up to assess the effects of the physical exercise protocol on neuroplasticity-related molecular markers.
Dopamine | Through study completion, an average of 1 year
  Dopamine (pg/ml) concentrations measured in urine will be measured in pre-intervention, post-intervention, at the midpoint of the intervention (2 months), and at the follow-up to assess the effects of the physical exercise protocol on reward-related molecular markers.

CONTACTS AND LOCATIONS:
Overall Officials: Sónia Sousa, PhD, Principal Investigator — Research Center in Psychology, School of Psychology, University of Minho